CLINICAL TRIAL: NCT06969846
Title: Direct Carotid Sinus Nerve Stimulation in Anesthetized Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan Baskin, Chief, Section of Otolaryngology-Head & Neck Surgery, Louis Stokes VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLINB0001; CLINB0001 (Other: VA Northeast Ohio Healthcare System)
Record Dates: First submitted 2025-04-04; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: HTN-Hypertension; Blood Pressure Management
Keywords: neuromodulation; hypertension; autonomic; electrode; implant
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Therapeutic Group (Experimental): Eligible patients were those scheduled to undergo elective surgical procedure that therapeutically indicated exposure of the carotid bifurcation and vascular sheath (e.g. carotid endarterectomy, neck dissection, or carotid tumor Resection) regardless of a HTN diagnosis. Exclusion criteria included disease states such as a history of stroke, or prior ipsilateral neck surgery or radiation treatment. Cardiovascular disease that precluded enrollment were diagnoses which independently increased surgical and anesthetic risk (American Society for Anesthesia Classification System).
  Interventions: Device: CSN electrode was implanted around tissue including CSN branches

INTERVENTIONS:
Device: CSN electrode was implanted around tissue including CSN branches — Using a novel surgical approach, a custom electrode was implanted around tissue including CSN branches in anesthetized adults. Following functional mapping, presumed baroafferent fibers were identified via response and stimulated. Outcome measures included change in systolic BP (SBP), diastolic BP (DBP), and heart rate (HR) during and after stimulation using multi-level modeling. Secondarily, dose dependency was examined.

SUMMARY:
Uncontrolled hypertension (HTN) is growing in incidence globally creating a critical need for alternative therapeutic strategies. Directly stimulating the carotid sinus nerve (CSN) is known to potentially reduce blood pressure (BP) but its clinical efficacy has not been consistently demonstrated with existing electrode technologies in humans.

We investigated the effect of acute direct CSN stimulation on BP and HR in anesthetized humans using an application-specific multi-contact electrode.

ELIGIBILITY:
Inclusion Criteria:

* . Eligible patients were those scheduled to undergo elective surgical procedure that therapeutically indicated exposure of the carotid bifurcation and vascular sheath (e.g. carotid endarterectomy, neck dissection, or carotid tumor Resection) regardless of a HTN diagnosis.

Exclusion Criteria:

* history of stroke
* prior ipsilateral neck surgery or radiation treatment
* Cardiovascular disease that precluded enrollment were diagnoses which independently increased surgical and anesthetic risk (American Society for Anesthesia Classification System).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Maximum drops and recovery in systolic blood pressure (SBP) as a result of carotid sinus nerve (CSN) stimulation | 1 hour
  The primary outcome was maximum drops and recovery in systolic blood pressure (SBP) as a function of carotid sinus nerve (CSN) stimulation as measured in mmHg. The maximum drop was calculated as the maximum change in SBP while stimulus was active, relative to the baseline value 30 seconds before starting stimulus. Maximum recovery was calculated as the largest change in SBP within 30 seconds of ending stimulus relative to the nadir in SBP (mmHg) during stimulation.

SECONDARY OUTCOMES:
The changes in blood pressure as a result of stimulation across all stimulation epochs | 1 hour
  The generalized drops and recoveries of systolic and diastolic blood pressure (SBP & DBP) measured in mmHg across all stimulation epochs as a function of CSN stimulation and stimulation withdrawal using the same timeframe as that used in the primary outcome.
The changes in heart rate as a result of stimulation across all stimulation epochs | 1 hour
  The generalized drops and recoveries in heart rate (HR) measured in beats per minute (BPM) as a result of stimulation and stimulation withdrawal across all stimulation epochs using the same time frame as #1.
Cumulative drops in SBP throughout entire stimulation session | 1 hour
  Individual patient cumulative drops in SBP (measured in mmHg) throughout the entire stimulation period/session were measured by pooling the baseline SBP values before the stimulation session began and the final SBP following the completion of the last stimulation epoch of the period.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Northeast Ohio Healthcare System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Majerus SJA, Pinault G, Tyler D, Dunning J, Schlesinger R, Heald E, Baskin JZ. Direct carotid sinus nerve stimulation in anesthetized human subjects. Sci Rep. 2025 Jul 21;15(1):26488. doi: 10.1038/s41598-025-10091-1. PMID 40691692